CLINICAL TRIAL: NCT04891887
Title: Diabetes Mellitus and microRNA as Risk Factors for Mild Cognitive Impairment: Impact of Life Style Modification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Science and Technology Development Fund (STDF) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15026
Record Dates: First submitted 2021-04-25; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes mellitus; Health education; Depression; Quality of life; Healthy life style; Cognitive function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Health Education; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Health education program
  Interventions: Behavioral: Health education program

INTERVENTIONS:
Behavioral: Health education program — Seven face to face sessions and group discussion health education sessions. Two prepared booklets were distributed to all attendants titled "Diabetes mellitus and how to control its complications" and "Mild cognitive impairment and how to prevent it".
  Lab results were discussed individually with each participant to discuss his adherence to the lifestyle modification program.
  Clinical follow-up and management with endocrinology and neurology specialists. Individualized Medical Nutrition. Participants were then counselled on healthy eating habits.
  Individualized biweekly follow-up scheme through mobile phone. A WhatsApp group was created for all participants to contact the research team whenever they have any inquiry concerning life style modifications. Through this group, 12 HE audio electronic messages were shared with participants.
  Final reassessment of clinical status and laboratory profile was carried out with participants who continued till the end of the study.

SUMMARY:
This is a 2-step study; 1st step was a cross sectional study carried out on 163 consecutive Type 2 Diabetes Mellitus (T2DM) patients employee attending outpatient clinics of the National Research Center (NRC), Egypt. A face-to-face interview was carried out to collect data about demographic data and medical history. Cognitive function assessment was carried out using Adenbrooke's Cognitive Examination III (ACE III) test and the Trail Making Test (TMT) which consists of two parts (A and B). Quality of life and depression were also assessed using Short Form-36 (SF-36) and Hamilton Depression Rating Scale (HRDS) questionnaires respectively. The second step was an interventional study for health education and life style modification. The main outcome measures were Fasting Blood Glucose (FBG), HbA1c, total blood cholesterol, HDL cholesterol, LDL cholesterol and triglycerides, oxidant and antioxidant (Malondialdehyde (MDA), glutathione peroxidase (GPx), glutathione reductase (GR)) which were assessed at baseline and reassessed after the intervention.

DETAILED DESCRIPTION:
The current study was carried out during the period from February 2016 to June 2019 on two steps.

1. First step (baseline assessment): It was a cross sectional study carried out on 163 Type 2 Diabetes Mellitus (T2DM) patients attending outpatient clinics at NRC. Patients were 65 males and 98 females; aged from 40 to 65 years. All patients were literate and were able to complete the tests of cognitive function. The exclusion criteria were T2DM patients with history of head trauma, stroke, transient ischemic attack, brain tumor, epilepsy, psychiatric disease, cardiac or liver failure and visual or hearing disabilities. Approval of NRC ethical committee was obtained with registration number 15131. Participants signed a written informed consent before being included in the study.

1.1 A face to face interview was carried out with all participants to collect data about demographics, medical history and cognitive function. Data included age, gender, level of education, and tobacco smoking. Detailed medical history of diabetes was taken from patients including age of diagnosis of diabetes, frequency of hypoglycemic attacks, type of treatment (insulin or oral hypoglycemic drug), history of hypertension, dyslipidemia or other diseases and medications taken. Any complaint suggestive for presence of sensory peripheral neuropathy such as tingling, burning pain or numbness in hands and feet was recorded. All studied participants were subjected to thorough clinical examination, systolic and diastolic blood pressure and anthropometric assessment (weight and height measurements).

1.2 Assessment of cognitive function with its domains was carried out using Adenbrooke's Cognitive Examination III (ACE III) test which assesses five cognitive domains: attention, memory, verbal fluency, language and visuospatial abilities. It is the most reliable and validated Arabic form cognitive scale and freely available to be applied. Objective mild cognitive impairment (MCI) was considered if ACE III score is less than 88. The Trail Making Test (TMT) was also used. TMT is one of the most widely used instruments in neuropsychological assessment as an indicator of speed of cognitive processing and executive functioning. It assesses attention, concentration, psychomotor speed, cognitive shifting and complex sequencing function by measuring the time required to connect a series of sequentially numbered and lettered circles. The test consists of two parts (A and B). The direct score of each part is represented by the time of completion of the tasks. Shorter time indicates better cognitive function.

1.3 Hamilton Rating Scale for Depression (HRSD) was used, it is one of the most widely used scales that objectively rate depression severity. The scale includes 17 items, each one is scored on a 3 or 5 points scale, with the final score indicative of the severity of the patient's depression. The classification of depression level was carried out depending on the National Institute for Health & Clinical Excellence of the United Kingdom (UK) (0-7 = Normal, 8-13 = Mild depression, 14-18 = Moderate depression, 19-22 = Severe depression and ≥ 23 = Very severe depression).

1.4 Assessment of health related quality of life (HRQOL) was carried out using Short Form-36 (SF-36) questionnaire. The questionnaire contains 36 items comprising eight domains of health status which are physical functioning (PF), role physical (RP), bodily pain (BP), general health perception GH), vitality (VT), social functioning (SF), role emotional (RE) and mental health (MH). Scoring of each domain is from 0 to 100, with a score of '100' as the best rating of health. The Arabic version of the questionnaire was used.

1.5 Assessment of T2DM patients' life style. Patients were given a designed questionnaire to assess their life style regarding nutritional habits, physical, social and mental activities and the opinion about the best way to motivate them for changing their lifestyle.

1.6 Baseline Laboratory analysis. Five ml blood sample was withdrawn under complete aseptic technique from each participant, after fasting for at least 10 hours at the beginning of the study. It was divided into dry plain and lavender ethylene diamine tetra acetic acid (EDTA) vacutainer tubes. Level of glycated hemoglobin (HbA1c) and total blood cholesterol were assessed using Olympus-au-400 chemistry auto-analyzer. Malondialdehyde (MDA) concentrations in serum was determined using ELISA kit based on the competitive binding enzyme immunoassay technique. Erythrocytes were examined for the enzymatic antioxidant activity of catalase, glutathione peroxidase (GPx) and glutathione reductase (GR).

1.7 For miRNAs expression analysis: Blood was drawn into special RNA preservation tubes; inverted 8-10 times, and then stored frozen at -80°C for further RNA extraction. RNA isolation and estimation of RNA quality was employed prior to initiating the characterization of miRNA expression. Only 1-10 nano grams of purified total RNA or equivalent was enough to reliably quantify the miRNAs of interest. The concentrations of miRNAs selected in this study was determined by the single target TaqMan miRNA quantitative Real Time (qRT) Polymerase Chain Reaction (PCR) assay (Applied Biosystems) in the plasma samples according to the manufacturer's instructions. A two-step protocol were applied which requires only reverse transcription with a miRNA-specific primer, followed by real-time PCR with TaqMan probes. The TaqMan MicroRNA Assays is a target-specific stem-loop structure reverse-transcription primer. The stem-loop accomplishes two goals: 1) specificity for only the mature miRNA target, and 2) formation of a Reverse Transcriptase (RT) primer/mature miRNA-chimera, extending the 5' end of the miRNA. RT reactions containing RNA samples, looped- primers, 1 X buffer, reverse transcriptase, and RNase inhibitor will be incubated for 30 min each, at 16°C and at 42°C. The resulting longer RT amplicon presents a template amenable to standard real-time PCR, using TaqMan assays. Then Real-time PCR was performed on Quant Studio 12 K Flex Real-Time PCR Instrument.

Second step (interventional trial): This step was an interventional study for health education and life style modification. It was carried out to Implementing the life style modification program on T2DM patients.

2.1 Designing two health educational booklets After identifying the T2DM participants' needs, the research team designed two health education booklets. The first booklet titled "Diabetes mellitus and how to control its complications". The booklet includes information about T2DM disease and, how it affects different body systems leading to Diabetes Mellitus (DM) complications. It includes also information on normal and abnormal level of fasting blood glucose and glycated hemoglobin (HbA1c). It demonstrates how to control and prevent DM complications, stressing on healthy nutrition and carbohydrate counting, physical activities, strict adherence to medical regimen and avoiding stress. The second booklet titled "Mild cognitive impairment and how to prevent" it includes information about definition of cognitive function, MCI and Alzheimer and its relation with T2DM and risk factors for cognitive impairment and how to control and improve cognitive function.

2.2 Patient education program implementation: Only 144 participants accepted the invitation to attend the health education (HE) sessions. The actual number who attended were only 121. The reasons for non-participation include: lack of interest and they refused commitment to the life style program.

2.2.1 Face to face and group discussion HE sessions to encourage life style modification: All the studied patients were invited to attend the HE sessions. Seven sessions were held at NRC over a period of nearly 2 months explaining the two designed booklets. HE lectures were presented by the public health team and a diabetic expert who shared in the group discussion to explain and answer the questions related to management of T2DM. HE program was provided for controlling DM, information about foods important to brain health and different intellectual games to improve their cognition.

2.2.2 Dissemination of Educational Materials The prepared booklets were distributed to all attendants. Participants were informed about the importance of these two booklets in improving their scientific information on T2DM and MCI.

2.2.3 Reassessment of laboratory analysis. Three ml of blood sample was withdrawn under complete aseptic technique from each participant, after fasting for at least 10 hours at the time of health education. It aimed to assess FBG, HbA1c and total blood cholesterol just before the intervention and were reassessed three months during the intervention to be an incentive for the patients as a monitoring the progress they attained due to life style modification. Each participant was asked to receive his laboratory results personally from the research team. This allowed to discuss the interpretation of his results and thus re-encourage or give him any needed advice to maintain his adherence to the lifestyle modification program.

2.2.4 Clinical follow-up and management were carried out by specialist in endocrinology and neurology depending on laboratory results and patient compliance.

2.2.5 Individualized Medical Nutrition program: Each participant was asked to complete a 3-day food diary. These were discussed with each participant individually through a face-to-face interview in order to advise and convince them to change their dietary habits . Every patient was taught how he can regulate his diet depending on the result of laboratory analysis and carbohydrate count.

2.2.6 Individualized biweekly follow-up scheme was also distributed as a guide for the targeted healthy behaviors needed to be changed which allowed self-monitoring of their achieved progress. Over a period of 6 months, the participants were followed up through mobile phone, using designed sheet, to assess patients' compliance and adherence to the life style modification program.

2.2.7 WhatsApp phone application group: The participants were welcomed to contact the research team whenever they had any inquiry concerning life style or treatment modifications. Through this group, 12 audio messages were recorded and distributed. These messages summarized the content of the booklet, to be an easily accessible way for the patients to help them follow the health education. Tips for healthy habits as well as exercises for mental activities were also uploaded to this group.

2.3.8 Final reassessment of clinical status and laboratory profile. Six months after recruitment, a face-to-face interview was carried out with the 98 participants who continued till the end of the study. They fulfilled a final sheet to assess their compliance to the program. ACE III test and TMT with its two parts A and B tests were reassessed with clinical, weight and blood pressure reassessment to evaluate the impact of the lifestyle modification program on cognitive function. Quality of life and depression were reassessed using SF-36 and HRDS questionnaires respectively. Laboratory analysis for the level of HbA1c, lipid profile, oxidant and antioxidant were reassessed after the intervention.

ELIGIBILITY:
Inclusion Criteria:

T2DM patients attending outpatient clinics of Medical Services Unit of the National Research Center (NRC).

Exclusion Criteria:

T2DM patients with history of head trauma, stroke, transient ischemic attack, brain tumor, epilepsy, psychiatric disease, cardiac or liver failure and visual or hearing disabilities

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months
  HbA1c
Cognitive function | 6 months
  Total score of Adenbrooke's Cognitive Examination III. Minimum value= 0, maximum value= 100 and higher scores mean a better outcome.
Depression | 6 months
  Hamilton Rating Scale for Depression score. Minimum value= 0, maximum value= 53 and higher scores mean a worse outcome.
Health related quality of life | 6 months
  Short Form-36 (SF-36) questionnaire score. Minimum value= 0, maximum value= 100 and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Malondialdehyde | 6 months
  Serum Malondialdehyde level
Glutathione Reductase | 6 months
  Erythrocyte Glutathione Reductase activity
Glutathione Peroxidase | 6 months
  Erythrocyte Glutathione Peroxidase activity
Total serum cholesterol | 6 months
  Total serum cholesterol level
LDL | 6 months
  serum LDL level
HDL | 6 months
  Serum HDL level
Triglycerides | 6 months
  Serum triglycerides level
Fasting blood glucose | 6 months
  Serum fasting blood glucose level
Healthy dietary intake | 6 months
  Questionnaire with the following items:
  1. Intake of fresh vegetables
  2. Intake of Dark green vegetable
  3. Intake of oats
  4. Healthy snacks
  5. Water intake
  6. Sugar intake
  7. Intake of yellow cheese
  8. Intake of Fried food
  9. Intake of margarine
  10. Intake of carbohydrate
  11. Intake of soft drinks
  12. Intake of sweets and deserts
  Minimum value= never or less than once/ month, maximum value= 2-3 time/ day
  For food items from 1-5, higher scores mean a better outcome and for food items from 6- 12, higher score means a worse outcome.
Physical activities | 6 months
  Physical activity questionnaire to assess the following:
  Light activities as walking
  Moderate activities
  Heavy activities
  Minimum value= 0, maximum value= 300 minutes/ week and higher scores mean a better outcome.
Social activity | 6 months
  Social activity questionnaire to assess the following:
  Going to restaurants and cafes
  Going to the club
  Participate in seminars in the mosque or church, social circles, and groups for entertainment
  Visiting relatives
  Going to museums, art galleries, theaters, cinemas, and concerts
  Minimum value= never or less than once/ month, maximum value= daily and higher scores mean a better outcome.
Mental activity | 6 months
  Mental activity questionnaire to assess daily practice of the following activities:
  Reading
  Listening to radio
  Playing Intellectual games
  Internet usage
  Minimum value= never or less than once/ month, maximum value= 4 hours/ day and higher score means a better outcome.
Trail Making Test | 6 months
  Trail Making Test
Medication compliance | 6 months
  Medication compliance was assessed by questionnaire include regularity of medication intake
  0=No 1=to some extent 2=sometimes 3=often 4=Always
  Higher score means a better outcome
Hypoglycemic attacks | 6 months
  The number of patients who complained of hypoglycaemic attacks
Body weight | 6 months
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: Iman I Salama, MD, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salama II, Sami SM, Salama SI, Abdel-Latif GA, Aboulghate A, Raslan HM, Mohsen A, Rasmy H, Ibrahim MH, Ganem MM, Abdelmohsen AM, El-Etreby LA, Ibrahim NA, Fouad WA, El-Deeb SE. Impact of lifestyle modification on glycemic control and cognitive function among Type II diabetes mellitus patients. Future Sci OA. 2023 Mar 9;9(1):FSO835. doi: 10.2144/fsoa-2022-0060. eCollection 2023 Jan. PMID 37006227